CLINICAL TRIAL: NCT07274319
Title: EFFICACY OF TRANSMUCOSAL MINIPLEITE STABILIZATION TECHNIQUE VERSUS INTRA-ARCH WIRE STABILIZATION TECHNIQUE FOR FIXATION OF SAGITTAL & PARA-SAGITTAL TYPES OF PALATAL FRACTURES IN TERMS OF INTRA-ARCH MOLAR DISTANCE & MAXILLO-MANDIBULAR MOLAR RELATION
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Services Institute of Medical Sciences, Pakistan (Other Government)
Responsible Party: Principal Investigator, Muhammad Hassan, Muhammad Hassan, Services Institute of Medical Sciences, Pakistan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB/2025/1699/SIMS
Record Dates: First submitted 2025-11-27; First posted 2025-12-10 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-11

CONDITIONS: Sagittal and Parasagittal Palatal Fracture
Keywords: sagittal palatal fracture; parasagittal palatal fracture

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intra arch wire stabilization (Active Comparator): . Technique for Intra-Arch Wire Stabilization:
  Anesthesia:
  Nasoendotracheal intubation combined with general anesthesia.
  Access via Surgery:
  The fracture line is identified.
  Positioning the Wire:
  Around the necks of the rear palatal teeth, stainless steel wires (often 26 or 28 gauge) are passed, commonly from molar to molar or second premolar to second premolar.
  To stabilize the segments and guarantee appropriate fracture reduction, the wires are crossed over the palate (transpalatal wiring).
  Alignment of Occlusal Space:
  To guarantee that the molar connection is preserved during tightening, temporary intermaxillary fixation (IMF) or occlusal guiding are employed.
  Occlusion is rechecked for correctness after stabilization.
  Care Following Surgery:
  oral hygiene guidelines, analgesics, and antibiotics. One to two weeks of a liquid-to-soft diet. Wires are removed in an outpatient setting and may stay in place for four to six weeks.
  Interventions: Procedure: intra arch wire stabilization technique
- Transmucosal Miniplate Stabilization (Experimental): Anesthesia:
  Nasoendotracheal intubation for general anesthesia.
  Adapting Plates:
  To fit the palatal curvature, a 1.5 or 2.0 mm titanium miniplate is molded.The plate is adapted over the fracture site and placed over the palate tissue.
  Fixing the Plate:
  The miniplate is attached to the palatal bone on each side of the fracture using miniscrews (4-6 mm).
  Intraoperative check-bite or temporary intermaxillary fixation are used to guide occlusion.
  Healing of Wounds:
  Because there is little disturbance, mucosal healing happens quickly.
  Care Following Surgery:
  standard regimen of analgesics and antibiotics. Rinses with chlorhexidine and soft diet. Unless exposed or symptomatic, the miniplate is often kept in place; a second surgery is not necessary unless it is necessary.
  Monitoring of Follow-Up and Outcomes:
  * Frequent follow-up appointments at 1, 2, 4, and 6 weeks.
  * intra-arch molar distance measurement with model analysis or digital calipers.
  * Using bite analysis or occlusal markers,
  Interventions: Procedure: Transmucosal Miniplate Stabilization

INTERVENTIONS:
Procedure: intra arch wire stabilization technique — Anesthesia:
  Nasoendotracheal intubation combined with general anesthesia.
  Access via Surgery:
  The fracture line is identified.
  Positioning the Wire:
  Around the necks of the rear palatal teeth, stainless steel wires (often 26 or 28 gauge) are passed, commonly from molar to molar or second premolar to second premolar.
  To stabilize the segments and guarantee appropriate fracture reduction, the wires are crossed over the palate (transpalatal wiring).
  Alignment of Occlusal Space:
  To guarantee that the molar connection is preserved during tightening, temporary intermaxillary fixation (IMF) or occlusal guiding are employed.
  Occlusion is rechecked for correctness after stabilization.
  Care Following Surgery:
  oral hygiene guidelines, analgesics, and antibiotics. One to two weeks of a liquid-to-soft diet. Wires are removed in an outpatient setting and may stay in place for four to six weeks.
  Arms: intra arch wire stabilization
Procedure: Transmucosal Miniplate Stabilization — Anesthesia:
  Nasoendotracheal intubation for general anesthesia.
  Adapting Plates:
  To fit the palatal curvature, a 1.5 or 2.0 mm titanium miniplate is molded.The plate is adapted over the fracture site and placed over the palate tissue.
  Fixing the Plate:
  The miniplate is attached to the palatal bone on each side of the fracture using miniscrews (4-6 mm).
  Intraoperative check-bite or temporary intermaxillary fixation are used to guide occlusion.
  Healing of Wounds:
  Because there is little disturbance, mucosal healing happens quickly.
  Care Following Surgery:
  standard regimen of analgesics and antibiotics. Rinses with chlorhexidine and soft diet. Unless exposed or symptomatic, the miniplate is often kept in place; a second surgery is not necessary unless it is necessary.
  Monitoring of Follow-Up and Outcomes:
  * Frequent follow-up appointments at 1, 2, 4, and 6 weeks.
  * intra-arch molar distance measurement with model analysis or digital calipers.
  * Using bite analysis or occlusal markers,
  Arms: Transmucosal Miniplate Stabilization

SUMMARY:
The purpose of this study is to reduce uncertainity around decision making regarding use of transmucosal miniplate stabilization technique in place of intra-arch wire stabilization technique to get better outcomes. It will help establish future guidelines for sagittal and para-sagittal types of palatal fracture treatment Under general anasthesia wires will be passed between molars of both sides for palatal fracture reduction or fracture will be reduced by applying plate at fracture site

DETAILED DESCRIPTION:
Patients who present to a tertiary care oral and maxillofacial surgery department with sagittal or parasagittal palatal fractures will have their data prospectively gathered. Participants will be randomized to either the intra-arch wire stabilization group or the transmucosal miniplate stabilization group after providing their informed consent and undergoing eligibility screening.

Details of the Surgical Procedure

1. Preoperative Assessment:

   A thorough clinical examination that includes a palatal integrity assessment and an occlusal evaluation.

   To verify the kind (sagittal or para-sagittal) and extent of a palatal fracture, radiological imaging (CT or 3D CBCT scans) will be used along with imprints of the mandible and maxilla for model analysis and preoperative anesthetic evaluation and preventative antibiotics.
2. Technique for Intra-Arch Wire Stabilization:

   Anesthesia:

   Nasoendotracheal intubation combined with general anesthesia.

   Access via Surgery:

   The fracture line is identified.

   Positioning the Wire:

   Around the necks of the rear palatal teeth, stainless steel wires (often 26 or 28 gauge) are passed, commonly from molar to molar or second premolar to second premolar.

   To stabilize the segments and guarantee appropriate fracture reduction, the wires are crossed over the palate (transpalatal wiring).

   Alignment of Occlusal Space:

   To guarantee that the molar connection is preserved during tightening, temporary intermaxillary fixation (IMF) or occlusal guiding are employed.

   Occlusion is rechecked for correctness after stabilization.

   Care Following Surgery:

   oral hygiene guidelines, analgesics, and antibiotics. One to two weeks of a liquid-to-soft diet. Wires are removed in an outpatient setting and may stay in place for four to six weeks.
3. Technique for Transmucosal Miniplate Stabilization:

Anesthesia:

Nasoendotracheal intubation for general anesthesia.

Adapting Plates:

To fit the palatal curvature, a 1.5 or 2.0 mm titanium miniplate is molded.The plate is adapted over the fracture site and placed over the palate tissue.

Fixing the Plate:

The miniplate is attached to the palatal bone on each side of the fracture using miniscrews (4-6 mm).

Intraoperative check-bite or temporary intermaxillary fixation are used to guide occlusion.

Healing of Wounds:

Because there is little disturbance, mucosal healing happens quickly.

Care Following Surgery:

standard regimen of analgesics and antibiotics. Rinses with chlorhexidine and soft diet. Unless exposed or symptomatic, the miniplate is often kept in place; a second surgery is not necessary unless it is necessary.

Monitoring of Follow-Up and Outcomes:

* Frequent follow-up appointments at 1, 2, 4, and 6 weeks.
* intra-arch molar distance measurement with model analysis or digital calipers.
* Using bite analysis or occlusal markers, the molar connection is evaluated.
* Using follow-up radiographs and clinical stability, fracture healing is evaluated.

Demographic information, trauma history, fracture classification (as verified by CT imaging), and the baseline intra-arch molar distance measured with digital calipers will all be included in the preoperative data. Standard occlusion classification will be used to clinically document baseline maxillo-mandibular molar relationships. Trained maxillofacial surgeons will carry out the designated surgical procedure according to a defined methodology.

Assessments for postoperative follow-up will be carried out at 1, 4, 8, and 12 weeks. Clinical assessments of occlusal stability, intra-arch molar distance measurements, postoperative complications, and the need for occlusal correction will all be recorded at each visit. To guarantee data quality, data will be entered using structured forms and checked for accuracy by a second reviewer.

ELIGIBILITY:
Inclusion Criteria:

* • Age ≥16 years

  * Both gender
  * CT scan confirmation of a sagittal or para-sagittal palatal fracture
  * Dentate patients whose first molars are intact

Exclusion Criteria:

* • Transverse or comminuted palatal fractures

  * Patients with edentulous teeth
  * Coagulopathies or serious systemic diseases
  * Patients who decline to follow up

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-09-01 (Estimated); Primary Completion 2027-02-28 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Maxillo-Mandibular Molar Relation | 4,8 and 12 weeks
  The upper and lower first molars' occlusal alignment is evaluated both clinically, to classify them as normal, mildly malocclusion, or severely malocclusion. Molar relationships are compared to Angle's classification by visual clinical assessment. The degree of malocclusion is determined by changes from before to after surgery.
Intra-Arch Molar Distance | 4, 8, and 12 weeks
  Before and after surgery, the inter-molar distance between the maxillary first molars was measured in millimeters using a digital caliper. measured using a digital caliper across the first molars' mesiobuccal cusp points before and after surgery; a change signifies collapse or widening of the arch.

SECONDARY OUTCOMES:
Occlusal Stability | 4, 8 and 12 weeks
  Over the course of eight to twelve weeks, the postoperative maintenance of the pre-injury occlusion without deviation or malalignment was evaluated. clinically assessed at every follow-up appointment (often at 4, 8, and 12 weeks); stability is verified if the occlusion doesn't alter in terms of functionality or appearance.

CONTACTS AND LOCATIONS:
Locations (1):
- Services Institute of Medical Sciences Lahore, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] 8. Bej A, Mishra S, Padhiary SK, Sahoo S, Kadam DR. A Prospective Study on Comparison of the Effectiveness of Transmucosal Plate and Intra-arch Wire Fixation in the Management of Palatal Fracture. Journal of Maxillofacial and Oral Surgery. 2025 Jun 8:1-6.
- [Result] Broaddus WC, Holloway KL, Winters CJ, Bullock MR, Graham RS, Mathern BE, Ward JD, Young HF. Titanium miniplates or stainless steel wire for cranial fixation: a prospective randomized comparison. J Neurosurg. 2002 Feb;96(2):244-7. doi: 10.3171/jns.2002.96.2.0244. PMID 11838797
- [Result] Cienfuegos R, Sierra E, Ortiz B, Fernandez G. Treatment of Palatal Fractures by Osteosynthesis with 2.0-mm Locking Plates as External Fixator. Craniomaxillofac Trauma Reconstr. 2010 Dec;3(4):223-30. doi: 10.1055/s-0030-1268519. PMID 22132261
- [Result] Giri KY, Sahu P, Rastogi S, Dandriyal R, Mall S, Singh AP, Indra B NP, Pratap Singh H. Bite Force Evaluation of Conventional Plating System Versus Locking Plating System for Mandibular Fracture. J Maxillofac Oral Surg. 2015 Dec;14(4):972-8. doi: 10.1007/s12663-015-0764-7. Epub 2015 Mar 10. PMID 26604472
- [Result] Silajiding K, Wusiman P, Yusufu B, Moming A. Three dimensional versus standard miniplate fixation in the management of mandibular fractures: A meta-analysis of randomized controlled trials. Kaohsiung J Med Sci. 2017 Sep;33(9):464-472. doi: 10.1016/j.kjms.2017.05.001. Epub 2017 Jun 29. PMID 28865605
- [Result] 3. Sharma D, Khan TA, Tripathi GM, Mishra A. Epidemiology, Pattern, and Management of Midsagittal and Parasagittal Palatal Fractures through Placement of Intra-arch Wire. Journal of Surgical Specialties and Rural Practice. 2023 Jan 1;4(1):28-32.
- [Result] Kumar U, Jain P. Sagittal Maxillary Fracture: Diagnosis and Management. Indian J Plast Surg. 2021 Aug 2;54(3):284-288. doi: 10.1055/s-0041-1729665. eCollection 2021 Sep. PMID 34667512
- [Result] Bhargava D, Thomas S, Pandey A. Reduction of Palatal Midline and Para-Midline Fractures Using Intra-arch Wire Fixation Versus Transmucosal Miniplate Stabilization: Prospective Randomized Clinical Study to Evaluate Postoperative Occlusion. J Maxillofac Oral Surg. 2018 Mar;17(1):71-74. doi: 10.1007/s12663-016-0980-9. Epub 2016 Oct 21. PMID 29382998